CLINICAL TRIAL: NCT07063303
Title: The Effect of Intermittent Feeding on Circadian Rhythm in Critical Illness
Brief Title: Circadian Rhythm in Critical Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atılım University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: atılımnut
Record Dates: First submitted 2025-05-06; First posted 2025-07-14 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Critical Illness
Keywords: critical illness; intermittent feeding; circadian rhythm
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: Patients admitted to the ICU who require enteral feeding for at least 10 days are randomly assigned to one of two groups:
  Intermittent Feeding Group, where enteral product is administered in scheduled intervals aligned with circadian rhythms.
  Continuous Feeding Group, following the standard ICU practice of continuous enteral nutrition.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent Feeding Group (Active Comparator): Patients receive enteral nutrition at scheduled intervals to align with circadian rhythms.
  Interventions: Other: Intermittent feeding
- Continuous Feeding Group (Active Comparator): Patients receive enteral nutrition continuously, following the standard ICU practice.
  Interventions: Other: Continuous feeding

INTERVENTIONS:
Other: Intermittent feeding — Feeding Frequency: Enteral nutrition will be provided every 4 to 6 hours via nasogastric tube.
  Feeding Volume: Each session will deliver 240 to 720 mL of enteral formula. Feeding Duration: Each feeding session will last approximately 20 to 60 minutes.
  Arms: Intermittent Feeding Group
Other: Continuous feeding — Feeding Frequency: Enteral nutrition will be administered continuously for 20 hours per day via nasogastric tube.
  Feeding Volume: The total daily volume will be divided evenly over the 20-hour infusion period, based on individual nutritional requirements.
  Feeding Duration: Each 24-hour cycle includes 20 hours of continuous feeding followed by a 4-hour rest period.
  Arms: Continuous Feeding Group

SUMMARY:
The goal of this clinical trial is to determine whether intermittent enteral feeding positively influences circadian rhythms in critically ill patients in intensive care units (ICUs). The main research questions are:

1. Does intermittent feeding improve circadian rhythms in ICU patients?
2. How does intermittent feeding affect metabolic markers and recovery outcomes? Researchers will compare intermittent feeding to continuous feeding, the current standard method, to assess its impact on circadian stability and patient health.

Participants will:

1. Receive intermittent enteral feeding or continuous enteral feeding for at least 10 days
2. Undergo blood sample collection at three time points daily (morning, afternoon, midnight) to analyze circadian gene expression and metabolic markers
3. Have their clinical condition, nutrition status, and recovery progress monitored throughout the study

DETAILED DESCRIPTION:
Circadian rhythms regulate various physiological processes over a 24-hour cycle, including sleep-wake patterns, digestion, blood pressure, and hormone secretion. These rhythms are primarily controlled by the suprachiasmatic nucleus in the hypothalamus and influenced by environmental cues (zeitgebers), such as light exposure and meal timing. Critically ill patients often experience circadian rhythm disruptions due to prolonged artificial lighting, sleep disturbances, and continuous feeding, which may negatively impact metabolic health, immune function, and recovery. Given the significance of meal timing in circadian regulation, intermittent feeding might serve as a therapeutic strategy to restore circadian balance in ICU patients.

This study is a prospective, randomized controlled trial and will be conducted at Ankara Training and Research Hospital's Anesthesia Intensive Care Unit. Ethical approval for the study has been obtained from Ankara Training and Research Hospital with decision number E-93471371-514.99-226714167.

Patients will be randomly assigned to one of two groups:

* Intermittent Feeding Group - enteral nutrition will be provided at scheduled intervals (4-6 times daily) for 20-60 minutes per session, aligning with circadian cycles. Light exposure will also be adjusted, ensuring darkness during night hours.
* Continuous Feeding Group - patients will receive standard continuous enteral nutrition, without specific adjustments for circadian rhythms.

Blood samples will be collected on Day 1 and Day 7 at 08:00, 16:00, and 00:00 to analyze Brain and muscle aryl hydrocarbon receptor nuclear antigen-1 (BMAL1), Cyrptochrome 1 (CRY1), and Period 2 (PER2) gene expression and biochemical markers. No invasive procedures will be performed beyond routine ICU care. Patients' medical history, nutritional status, and clinical parameters will be recorded by using Acute Physiology and Chronic Health Evaluation II (APACHE II) Score, Sequential Organ Failure Assessment (SOFA) Score, Nutrition Risk in Critically ill (NUTRIC) Score and Global Leadership Initiative on Malnutrition (GLIM) Criteria.

ELIGIBILITY:
Inclusion Criteria:

* ICU admission for enteral feeding via a gastric tube
* Expected ≥10 days of enteral nutrition
* Age ≥18 years

Exclusion Criteria:

* Age <18 years
* Pregnancy
* Gastrointestinal surgery or diseases
* Tolerance issues with enteral feeding
* Parenteral feeding requirement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-09-29 (Actual); Study Completion 2025-09-29 (Actual)

PRIMARY OUTCOMES:
BMAL1 mRNA Expression Level | From randomization to the end of intervention (7 days)
  To evaluate the circadian rhythm in critically ill patients, BMAL1 gene expression will be measured using blood samples collected at 08:00, 16:00, and 00:00 on Day 1 and Day 7
CRY1 mRNA Expression Level | From randomization to the end of intervention (7 days)
  To evaluate the circadian rhythm in critically ill patients, CRY1 gene expression will be measured using blood samples collected at 08:00, 16:00, and 00:00 on Day 1 and Day 7
PER2 mRNA Expression Level | From randomization to the end of intervention (7 days)
  To evaluate the circadian rhythm in critically ill patients, PER2 gene expression will be measured using blood samples collected at 08:00, 16:00, and 00:00 on Day 1 and Day 7

SECONDARY OUTCOMES:
Fasting Glucose Level | From randomization to Day 7
  This parameter will be analyzed from blood samples collected on the first and seventh days after randomization. Unit of Measure: mg/dL
C-reactive protein (CRP) | From randomization to Day 7
  This parameter will be analyzed from blood samples collected on the first and seventh days after randomization. Unit of Measure: mg/L
Lactate Level | From randomization to Day 7
  This parameter will be analyzed from blood samples collected on the first and seventh days after randomization. Unit of Measure: mmol/L
Creatinine Level | From randomization to Day 7
  This parameter will be analyzed from blood samples collected on the first and seventh days after randomization. Unit of Measure: mg/dL
Bicarbonate Level | From randomization to Day 7
  This parameter will be analyzed from blood samples collected on the first and seventh days after randomization. Unit of Measure: mmol/L
White Blood Cell (WBC) Count | From randomization to Day 7
  WBC count (x10³/μL) will be analyzed from blood samples collected on the first and seventh days after randomization.
Lymphocyte Count | From randomization to Day 7
  Lymphocyte Count (x10³/μL) will be analyzed from blood samples collected on the first and seventh days after randomization.
Neutrophil Count | From randomization to Day 7
  Neutrophil Count (x10³/μL) will be analyzed from blood samples collected on the first and seventh days after randomization.
Hemoglobin Level | From randomization to Day 7
  Hemoglobin Level will be analyzed from blood samples collected on the first and seventh days after randomization. Unit of measure: g/dL
Platelet Count | From randomization to Day 7
  Platelet Count (x10³/μL) will be analyzed from blood samples collected on the first and seventh days after randomization.
Aspartate aminotransferase (AST) Levels | From randomization to Day 7
  Aspartate aminotransferase (AST) (U/L) levels will be analyzed from blood samples collected on the first and seventh days after randomization.
Alanine aminotransferase (ALT) Levels | From randomization to Day 7
  Alanine aminotransferase (ALT) (U/L) levels will be analyzed from blood samples collected on the first and seventh days after randomization.
Gamma glutamyl transferase (GGT) Levels | From randomization to Day 7
  Gamma glutamyl transferase (GGT) (U/L) levels will be analyzed from blood samples collected on the first and seventh days after randomization.
Blood Urea Nitrogen (BUN) Levels | From randomization to Day 7
  Blood Urea Nitrogen (BUN) (mg/dL) levels will be analyzed from blood samples collected on the first and seventh days after randomization.
Sodium Levels | From randomization to Day 7
  Sodium (mmol/L) levels will be analyzed from blood samples collected on the first and seventh days after randomization.
Potassium Levels | From randomization to Day 7
  Potassium (mmol/L) levels will be analyzed from blood samples collected on the first and seventh days after randomization.
Acute Physiology and Chronic Health Evaluation II (APACHE-II) Score | First day of admission to the ICU
  The APACHE II score is a clinical tool used in intensive care units to assess the severity of a patient's illness and estimate the risk of hospital mortality. It is calculated based on physiological measurements, age, and chronic health conditions. Higher scores indicate more severe illness and a greater risk of death.
  Unit of Measure: Score (0-71 scale) Interpretation: Higher scores correspond to increased severity and mortality risk.
Sequential Organ Failure Assessment (SOFA) Score | First day of admission to the ICU
  The SOFA score evaluates the function of six organ systems-respiratory, cardiovascular, hepatic, coagulation, renal, and neurological-in critically ill patients. It is used to monitor the extent of organ dysfunction and predict clinical outcomes in the intensive care unit (ICU).
  Unit of Measure: Score (0-24 scale) Interpretation: Higher scores indicate greater organ dysfunction and worse prognosis.
Nutrition Risk in Critically ill (NUTRIC) Score | First day of admission to the ICU
  The NUTRIC score is a screening tool designed to identify critically ill patients at high nutritional risk. It incorporates factors such as age, severity of illness, comorbidities, and inflammation to guide nutritional interventions in the intensive care unit (ICU).
  Unit of Measure: Score (0-10 scale) Interpretation: Higher scores indicate greater nutritional risk.
Global Leadership Initiative on Malnutrition (GLIM) Criteria | First day of admission to the ICU
  The GLIM criteria provide a standardized framework to diagnose malnutrition based on a combination of phenotypic criteria (including weight loss, low BMI, and reduced muscle mass) and etiologic criteria (such as reduced food intake or disease burden/inflammation). These criteria are used across clinical settings to identify malnutrition and grade its severity.
  Unit of Measure: Categorical (e.g., malnutrition diagnosed: yes/no; severity graded as mild, moderate, or severe)

CONTACTS AND LOCATIONS:
Overall Officials: Aslı Akyol Mutlu, Prof., Study Chair — Hacettepe University
Locations (1):
- Ankara Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) from this study due to ethical considerations and restrictions related to patient confidentiality in the ICU setting.

REFERENCES:
- [Background] Sagun E, Akyol A, Kaymak C. Chrononutrition in Critical Illness. Nutr Rev. 2025 Mar 1;83(3):e1146-e1157. doi: 10.1093/nutrit/nuae078. PMID 38904422
- [Background] Theilla M, Rattanachaiwong S, Kagan I, Rigler M, Bendavid I, Singer P. Validation of GLIM malnutrition criteria for diagnosis of malnutrition in ICU patients: An observational study. Clin Nutr. 2021 May;40(5):3578-3584. doi: 10.1016/j.clnu.2020.12.021. Epub 2020 Dec 29. PMID 33413910
- [Background] Jensen GL, Cederholm T, Correia MITD, Gonzalez MC, Fukushima R, Higashiguchi T, de Baptista GA, Barazzoni R, Blaauw R, Coats AJS, Crivelli A, Evans DC, Gramlich L, Fuchs-Tarlovsky V, Keller H, Llido L, Malone A, Mogensen KM, Morley JE, Muscaritoli M, Nyulasi I, Pirlich M, Pisprasert V, de van der Schueren M, Siltharm S, Singer P, Tappenden KA, Velasco N, Waitzberg DL, Yamwong P, Yu J, Compher C, Van Gossum A. GLIM Criteria for the Diagnosis of Malnutrition: A Consensus Report From the Global Clinical Nutrition Community. JPEN J Parenter Enteral Nutr. 2019 Jan;43(1):32-40. doi: 10.1002/jpen.1440. Epub 2018 Sep 2. PMID 30175461
- [Background] Van Dyck L, Vanhorebeek I, Wilmer A, Schrijvers A, Derese I, Mebis L, Wouters PJ, Van den Berghe G, Gunst J, Casaer MP. Towards a fasting-mimicking diet for critically ill patients: the pilot randomized crossover ICU-FM-1 study. Crit Care. 2020 May 24;24(1):249. doi: 10.1186/s13054-020-02987-3. PMID 32448392
- [Background] Kouw IWK, Heilbronn LK, van Zanten ARH. Intermittent feeding and circadian rhythm in critical illness. Curr Opin Crit Care. 2022 Aug 1;28(4):381-388. doi: 10.1097/MCC.0000000000000960. Epub 2022 Jul 5. PMID 35797531
- [Background] Sunderram J, Sofou S, Kamisoglu K, Karantza V, Androulakis IP. Time-restricted feeding and the realignment of biological rhythms: translational opportunities and challenges. J Transl Med. 2014 Mar 28;12:79. doi: 10.1186/1479-5876-12-79. PMID 24674294
- [Background] Ren CJ, Yao B, Tuo M, Lin H, Wan XY, Pang XF. Comparison of sequential feeding and continuous feeding on the blood glucose of critically ill patients: a non-inferiority randomized controlled trial. Chin Med J (Engl). 2021 Jul 20;134(14):1695-1700. doi: 10.1097/CM9.0000000000001684. PMID 34397596
- [Background] Dong J, Liu R, Li L, Yao L. [Effects of intermittent feeding and continuous feeding on muscle atrophy and nutritional status in critically ill patients]. Zhonghua Wei Zhong Bing Ji Jiu Yi Xue. 2021 Jul;33(7):844-848. doi: 10.3760/cma.j.cn121430-20210408-00517. Chinese. PMID 34412755
- [Background] Ichimaru S. Methods of Enteral Nutrition Administration in Critically Ill Patients: Continuous, Cyclic, Intermittent, and Bolus Feeding. Nutr Clin Pract. 2018 Dec;33(6):790-795. doi: 10.1002/ncp.10105. Epub 2018 Jun 20. PMID 29924423
- [Background] Jobanputra AM, Scharf MT, Androulakis IP, Sunderram J. Circadian Disruption in Critical Illness. Front Neurol. 2020 Aug 11;11:820. doi: 10.3389/fneur.2020.00820. eCollection 2020. PMID 32849248
- [Background] Acuna-Fernandez C, Marin JS, Diaz-Casado ME, Rusanova I, Darias-Delbey B, Perez-Guillama L, Florido-Ruiz J, Acuna-Castroviejo D. Daily Changes in the Expression of Clock Genes in Sepsis and Their Relation with Sepsis Outcome and Urinary Excretion of 6-Sulfatoximelatonin. Shock. 2020 May;53(5):550-559. doi: 10.1097/SHK.0000000000001433. PMID 31403491
- [Background] Diaz E, Diaz I, Del Busto C, Escudero D, Perez S. Clock Genes Disruption in the Intensive Care Unit. J Intensive Care Med. 2020 Dec;35(12):1497-1504. doi: 10.1177/0885066619876572. Epub 2019 Sep 11. PMID 31510864
- [Background] Maas MB, Iwanaszko M, Lizza BD, Reid KJ, Braun RI, Zee PC. Circadian Gene Expression Rhythms During Critical Illness. Crit Care Med. 2020 Dec;48(12):e1294-e1299. doi: 10.1097/CCM.0000000000004697. PMID 33031153
- [Background] Beyer SE, Salgado C, Garcao I, Celi LA, Vieira S. Circadian rhythm in critically ill patients: Insights from the eICU Database. Cardiovasc Digit Health J. 2021 Feb 17;2(2):118-125. doi: 10.1016/j.cvdhj.2021.01.004. eCollection 2021 Apr. PMID 35265899
- [Background] Coiffard B, Diallo AB, Culver A, Mezouar S, Hammad E, Vigne C, Nicolino-Brunet C, Dignat-George F, Baumstarck K, Boucekine M, Leone M, Mege JL. Circadian Rhythm Disruption and Sepsis in Severe Trauma Patients. Shock. 2019 Jul;52(1):29-36. doi: 10.1097/SHK.0000000000001241. PMID 30074979
- [Background] Neves AR, Albuquerque T, Quintela T, Costa D. Circadian rhythm and disease: Relationship, new insights, and future perspectives. J Cell Physiol. 2022 Aug;237(8):3239-3256. doi: 10.1002/jcp.30815. Epub 2022 Jun 13. PMID 35696609